CLINICAL TRIAL: NCT00154492
Title: Effectiveness and Safety of Use of NovoSeven® in the Treatment of Active Variceal Bleeding in Patients With Advanced Cirrhosis
Brief Title: Use of NovoSeven® in Active Variceal Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7LIVER-1533
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cirrhosis
Keywords: Active variceal bleeding in patients with advanced cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Asia and Europe. The trial is planned to investigate the effectiveness and safety of NovoSeven® in patients with advanced cirrhosis and active variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Variceal bleeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2004-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Treatment failure | Within 5 days after first trial product administration

SECONDARY OUTCOMES:
Mortality
Rebleeding
Control of acute bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- Novo Nordisk Investigational Site, Vienna, Austria
- Czechia (2):
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Prague
- Novo Nordisk Investigational Site, Aarhus, Denmark
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (12):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Clichy
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Limoges
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Villejuif
- Germany (6):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Ulm
- Novo Nordisk Investigational Site, Shatin, Hong Kong
- Italy (3):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Palermo
- Poland (3):
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Warsaw
- Spain (5):
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Majadahonda
- Novo Nordisk Investigational Site, Taipei, Taiwan
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com